CLINICAL TRIAL: NCT03590145
Title: Reliability of the Doha Agreement Classification in the Clinical Diagnosis of Groin Pain in Athletes - an Inter-examiner Reproducibility Study.
Brief Title: Reliability of the Doha Agreement Classification of Groin Pain
Status: Completed | Type: Observational
Sponsor: Aspetar (Other)
Collaborators: University College Dublin (Other)
Responsible Party: Principal Investigator, Andreas Serner, Clinical Research Scientist, Aspetar
Other Study IDs: Aspetar
Record Dates: First submitted 2018-06-26; First posted 2018-07-18 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Groin Injury; Hip Pain Chronic; Adductor Tendinitis; Inguinal Hernia; Iliopsoas Syndrome
Keywords: Groin pain; Adductor-related; Inguinal-related; Pubic-related; Iliopsoas-related; Hip-related
MeSH Terms: conditions — Hernia, Inguinal | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Qatari athletes: Participants meeting general inclusion criteria.
  Interventions: Diagnostic Test: Clinical examination

INTERVENTIONS:
Diagnostic Test: Clinical examination — Standardized clinical examination consisting of pain provocation test, including palpation, muscle resistance and stretch test.

SUMMARY:
This study will investigate the reproducibility of a clinical diagnostic classification system for groin pain between two different examiners.

DETAILED DESCRIPTION:
Groin pain is prevalent in field and court sport athletes. It is particularly prevalent in soccer, Gaelic football and rugby union. The wide variety of possible injuries in numerous anatomical structures and high prevalence of "abnormal imaging findings" in asymptomatic athletes contribute to the complexity. Heterogeneous taxonomy of groin injuries in athletes adds further to the confusion. Clinical practice is challenging with clinicians using differing groin pain terminology, where even the same term can have multiple interpretations. A recent systematic review on the treatment of groin pain in athletes included 72 studies, in which 33 different diagnostic terms were used. The "Doha agreement meeting on terminology and definitions in groin pain in athletes" was convened to attempt to resolve this problem. The Doha agreement meeting on terminology and definitions in groin pain in athletes reached a consensus on a clinically based taxonomy using three major categories. These definitions and terminology are based on history and physical examination to categorize athletes, making it simple and suitable for both clinical practice and research.

The purpose of this study is therefore to investigate the inter-examiner reliability of the "Doha agreement meeting on terminology and definitions in groin pain in athletes." The study will be performed at a Sports Medicine Hospital in Qatar.

Prior to the clinical examination participants will be requested to complete the Copenhagen Hip and Groin Outcome Score (HAGOS). This is a patient-reported outcome measure, which quantifies a patient's current subjective perception of their hip and groin pain within the last week on six subscales, each with a score between 0 and 100. Additionally, participants will be requested to complete the Oslo Sports Trauma Research Center (OSTRC) overuse injury questionnaire with a focus on groin problems within the last week.

A standardized clinical examination will be performed. Palpation, resistance testing and stretching of affected muscle groups are used to categorize athletes into defined clinical entities. The pain reported by the athlete during the tests should also be felt in the affected structure. For example, in adductor-related groin pain, the pain on resisted adduction testing should reproduce the athlete's recognizable pain in the adductors. Pain felt in a different location-for example, the inguinal region on resisted adduction testing-would not signify adductor-related groin pain.

Statistical analyses Cohen's Kappa statistic (κ) is used to signify agreement between clinicians. Agreement was considered almost perfect if κ=0.81-1.00, moderate κ=0.41-0.60, substantial κ=0.61-0.80, fair κ=0.21-0.40, slight κ=0-0.20, and poor if κ<0. In addition, absolute agreement, prevalence, and bias index will be calculated. Statistical analyses will be performed using SPSS software.

Sample size With two examiners at each site, an expected Kappa of at least 0.8 with a lower limit of a 95% confidence interval of 0.4, and an expected prevalence between 0.3-0.7 for the three expected main defined clinical entities (adductor-related, inguinal-related, and iliopsoas-related groin pain), assuming no bias between examiners, the required sample size is determined to be 48 using a 2-tailed test. As pubic-related and hip-related groin pain is expected to be less frequent, a lower limit confidence interval of 0 for these entities is accepted, which in a 1-tailed test, maintaining an expected kappa of 0.8, requires a sample of only 10 participants. Thus 48 participants will be included.

ELIGIBILITY:
Inclusion Criteria:

* adult (˃18y) male individuals regularly participating in recreational or elite sports activity (≥once/week).
* current primary complaint of hip and/or groin pain of a non-acute onset that worsens on exercise, or of acute onset, which has not recovered and become longstanding (˃6w).

Exclusion Criteria:

* any prior assessment or treatment from one of the examiners for the same complaints.
* fractures or acute injuries with severe pain were it would be unethical to examine the athlete twice.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult male individuals regularly participating in recreational or elite sports activity (≥once/week) with a current primary complaint of hip and/or groin pain of a non-acute onset that worsens on exercise, or of acute onset, which has not recovered and become longstanding (˃6w).
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Clinical entity | Oct 2017 - June 2019
  Patients are diagnosed with one or multiple clinical entities:
  "Adductor-related" (adductor tenderness AND pain on resisted adduction testing), "Pubic-related" (local tenderness of the pubic symphysis and the immediately adjacent bone), "Iliopsoas-related" (iliopsoas tenderness AND more likely with pain on resisted hip flexion AND/OR pain on stretching of the iliopsoas), "Inguinal-related" (pain location in the inguinal canal region AND tenderness of the inguinal canal. No palpable inguinal hernia. More likely if the pain is aggravated with resistance testing of the abdominal muscles OR on Valsalva/cough/sneeze), or "Hip-related" (clinical suspicion, either through history or clinical examination. Specific diagnosis will require further investigations and will not be included in this study), or "Other" (any cause of groin pain which cannot be included with in the specified clinical entities).

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Tol, PhD, Study Director — Aspetar Orthopaedic and Sports Medicine Hospital
Locations (1):
- Aspetar Orthopaedic and Sports Medicine Hospital, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided
There is currently no plan of sharing individual participant data; however, upon reasonable request, anonymized data can be made available for interested parties.

REFERENCES:
- [Background] Branci S, Thorborg K, Nielsen MB, Holmich P. Radiological findings in symphyseal and adductor-related groin pain in athletes: a critical review of the literature. Br J Sports Med. 2013 Jul;47(10):611-9. doi: 10.1136/bjsports-2012-091905. Epub 2013 Feb 12. PMID 23403531
- [Background] Serner A, van Eijck CH, Beumer BR, Holmich P, Weir A, de Vos RJ. Study quality on groin injury management remains low: a systematic review on treatment of groin pain in athletes. Br J Sports Med. 2015 Jun;49(12):813. doi: 10.1136/bjsports-2014-094256. Epub 2015 Jan 29. PMID 25633830
- [Background] Thorborg K, Holmich P, Christensen R, Petersen J, Roos EM. The Copenhagen Hip and Groin Outcome Score (HAGOS): development and validation according to the COSMIN checklist. Br J Sports Med. 2011 May;45(6):478-91. doi: 10.1136/bjsm.2010.080937. PMID 21478502
- [Background] Clarsen B, Myklebust G, Bahr R. Development and validation of a new method for the registration of overuse injuries in sports injury epidemiology: the Oslo Sports Trauma Research Centre (OSTRC) overuse injury questionnaire. Br J Sports Med. 2013 May;47(8):495-502. doi: 10.1136/bjsports-2012-091524. Epub 2012 Oct 4. PMID 23038786
- [Background] Weir A, Brukner P, Delahunt E, Ekstrand J, Griffin D, Khan KM, Lovell G, Meyers WC, Muschaweck U, Orchard J, Paajanen H, Philippon M, Reboul G, Robinson P, Schache AG, Schilders E, Serner A, Silvers H, Thorborg K, Tyler T, Verrall G, de Vos RJ, Vuckovic Z, Holmich P. Doha agreement meeting on terminology and definitions in groin pain in athletes. Br J Sports Med. 2015 Jun;49(12):768-74. doi: 10.1136/bjsports-2015-094869. PMID 26031643
- [Background] Landis JR, Koch GG. The measurement of observer agreement for categorical data. Biometrics. 1977 Mar;33(1):159-74. PMID 843571
- [Background] Taylor R, Vuckovic Z, Mosler A, Agricola R, Otten R, Jacobsen P, Holmich P, Weir A. Multidisciplinary Assessment of 100 Athletes With Groin Pain Using the Doha Agreement: High Prevalence of Adductor-Related Groin Pain in Conjunction With Multiple Causes. Clin J Sport Med. 2018 Jul;28(4):364-369. doi: 10.1097/JSM.0000000000000469. PMID 28654441
- [Background] Sim J, Wright CC. The kappa statistic in reliability studies: use, interpretation, and sample size requirements. Phys Ther. 2005 Mar;85(3):257-68. PMID 15733050